CLINICAL TRIAL: NCT07339956
Title: Yiwei Jiaohuang Ointment for Gastrointestinal Bleeding Associated With Oral Antithrombotic Agents: A Randomized Controlled Trial
Brief Title: Yiwei Jiaohuang Ointment for Gastrointestinal Bleeding Associated With Oral Antithrombotic Agents
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jie, Zhang, Attending Physician, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-NHLHCRF-PY-31
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Gastrointestinal Bleeding
Keywords: Antithrombotic therapy; Traditional Chinese Medicine
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Drug: A Chinese herb formula--Yiwei Jiaohuang Onitment; Drug: Rabeprazole Enteric-Coated Tablets
- Control (Active Comparator)
  Interventions: Drug: Rabeprazole Enteric-Coated Tablets

INTERVENTIONS:
Drug: A Chinese herb formula--Yiwei Jiaohuang Onitment — Yiwei Jiaohuang Onitment consists of four Chinese herbs: 3g of Duyiwei（Lamiophlomis Herb）, 3g of raw Da Huang(Rhubarb Root and Rhizome (Unprocessed)), 6g of Bai Ji(Bletilla Rhizome) and 10g of Ejiao (donkey-hide gelatin). Prepared as ointment, patients should take one dose daily in the morning on an empty stomach for 2 weeks.
  Arms: Intervention
Drug: Rabeprazole Enteric-Coated Tablets — Rabeprazole Enteric-Coated Tablets10mg once a day for 2 weeks

SUMMARY:
The goal of this clinical trial is to evaluate the clinical efficacy and safety of YiWei Jiaohuang Ointment in treating gastrointestinal bleeding associated with oral antithrombotic therapy. The main question it aims to answer is:

Does Yiwei JiaoHuang Ointment accelerate the conversion to negative results in fecal occult blood tests among patients with gastrointestinal bleeding associated with antithrombotic therapy? Researchers will compare use rabeprazole alone as routine therapy to see if Yiwei JiaoHuang Ointment can accelerate the conversion to negative results in fecal occult blood tests.

Participants will ： Take Yiwei JiaoHuang Ointment every day for 2 weeks. Return to the hospital for a fecal occult blood test after 3 days, 1 week, and 2 weeks of medication.

ELIGIBILITY:
Inclusion Criteria:

* Oral therapy with at least one antiplatelet or anticoagulant agent, including: aspirin, clopidogrel, ticagrelor, prasugrel, warfarin, rivaroxaban, apixaban, edoxaban, dabigatran, etc.;
* BARC stage 1 or 2;
* Traditional Chinese Medicine pattern identified as phlegm-heat and blood stasis obstruction syndrome;
* Age 18-90 years;
* Signed informed consent.

Exclusion Criteria:

* Patients with gastrointestinal bleeding resulting in hemoglobin levels <20 g/L and/or requiring hospitalization;
* Gastrointestinal malignancies;
* Cases where the source of occult blood cannot be distinguished, such as fresh bleeding from hemorrhoids;
* Concurrent use of hemostatic traditional Chinese medicine preparations like Yunnan Baiyao;
* Significant liver or kidney dysfunction, with ALT, AST, or serum creatinine exceeding three times the upper limit of normal;
* Pregnant women, women planning pregnancy, or lactating women;
* Individuals deemed unsuitable for this clinical trial by the investigator.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
The rate of negative fecal occult blood test results in the two groups of patients after 2 weeks of intervention. | two weeks of intervention

SECONDARY OUTCOMES:
Time required for fecal occult blood to turn negative in two groups of patients. | two weeks of intervention
The rate of negative fecal occult blood test results in the two groups of patients after 3 days of intervention. | 3 days of intervention
The rate of negative fecal occult blood test results in the two groups of patients after one week of intervention. | one week of intervention
Changes in hemoglobin levels in two groups of patients after 2 weeks of intervention. | two weeks of intervention

OTHER OUTCOMES:
Changes in Gut Microbiota Before and After Treatment in Two Groups of Patients | two weeks of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No